CLINICAL TRIAL: NCT05811195
Title: Comparison of Two Prophylactic Photobiomodulation Protocols in Chemoinduced Oral Mucositis in Pediatric and Adolescent Oncology Patients: a Randomized, Controlled, Blinded Clinical Trial
Brief Title: Comparison of Prophylactic Photobiomodulation Protocols in Chemoinduced Oral Mucositis in Oncology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital A.C. Camargo (Other)
Responsible Party: Principal Investigator, Manoela Domingues Martins, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBM and MO IN CHEMIOINDUCED
Record Dates: First submitted 2023-03-17; First posted 2023-04-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Oral Mucositis; Chemotherapeutic Toxicity; Childhood Cancer
MeSH Terms: conditions — Stomatitis; Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be allocated and randomized into 2 groups: Group I: PBMI (n=17) photobiomodulation intra oral low potency laser and Group II: PBME (n=17) photobiomodulation with high potency extraoral unfocoused laser with 1W.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assesor will not know the laser protocol of each patient (single blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intraoral photobiomodulation (PBMI) (Active Comparator): Intraoral application: A low-power laser (Diode Semiconductor, Duo, MMOptics Ltda, São Carlos, SP, Brazil) with a wavelength of 660 nm (red). Four anatomical areas will be irradiated perpendicularly in oral mucosa through several anatomical points with a distance of 1 cm approximately between them in order to cover the largest area per cm² in each region.
  Application points:
  * Jugal mucosa: 4 points for each side: upper and lower internal buccal vestibule, (8 points).
  * Jugal mucosa for younger children 2 points internal buccal vestibule in the center - each side (4 points)
  * Tongue: 2 points on right and left lateral border and 1 point on right and left belly (6 points)
  * Oral floor: (2 points).
  * Upper and lower lips: 2 points on upper inner labial mucosa, 2 points on lower inner labial mucosa (4 points).
  * Soft palate: right and left sides (2 points)
  Interventions: Device: Diode Semiconductor, Duo
- Extraoral photobiomodulation (PBME) (Active Comparator): A gallium-aluminum arsenide diode laser (Gemini® manufactured by Azena Medical, LLC, distributed by Ultradent Products, Inc.) with double wavelength 810 + 980 nm. The equipment will be programmed with 1 W of power.
  * 4 points - on each side of the face (2 on the right 2 on the left);
  * 2 points - on each side of the face: for younger children 1 point will be performed on each side of the face (1 on the right, 1 on the left)
  * 1 point on the lip; patients with sealed lips being able to cover both the upper and lower lip;
  * 5 points in the neck region (2 in right submandibular space and 2 in left submandibular space and submental space in the midline).
  * 3 points in the neck region for younger children (1 in right submandibular space and 1 in left submandibular space and submental space in the midline)
  Interventions: Device: Gemini laser

INTERVENTIONS:
Device: Diode Semiconductor, Duo — Intraoral photobiomodulation therapy (660nm, 3s/point, 10J/cm²) for the management for the oral mucositis in pediatric patients. Mainly in the decrease of oral mucositis rates severity, healing of the ulcers of OM. The results obtained will be compared with the other group.
  Arms: Intraoral photobiomodulation (PBMI)
Device: Gemini laser — Extraoral photobiomodulation therapy (810 + 980 nm, 20s/point, 4.07J/cm²) for the management for the oral mucositis in pediatric patients. Mainly in the decrease of oral mucositis rates severity, healing of the ulcers of OM. The results obtained will be compared with the other group.
  Arms: Extraoral photobiomodulation (PBME)

SUMMARY:
Childhood cancers represent less than 1% of the malignant diseases diagnosed worldwide. Treatment modalities for childhood malignancies will differ depending on the diagnosis. The main treatments may include chemotherapy (QT), radiation therapy (RT), and surgery. The toxicity caused by QT and RT generates adverse effects in the mouth, among them oral mucositis (MO). MO is damage that occurs to the oral mucosa and these lesions are extremely painful, uncomfortable, and cause great morbidity for patients. The main treatment of MO is intraoral photobiomodulation therapy (TBMI), this therapy has been widely used, reducing the severity and pain of MO in patients. The use of extraoral photobiomodulation therapy (TFBME) has been employed in some recent studies and has shown efficacy for reducing and improving the severity of OM. The present study aims to compare the effect of two protocols of photobiomodulation therapy (TFBM) using intraoral and extraoral low power laser in the prevention and treatment of OM in pediatric oncology patients receiving treatment with high dose metrotexate (MTX-HD) and its chemotherapy combinations. Initially, 34 pediatric and adolescent oncology patients receiving intravenous (IV) QT from risk protocols will be selected. Participants will be allocated into 2 groups: Group I: TFBMI (n=17) and Group II: TFBME (n=17). The study will be conducted by a dental surgeon who will perform the initial assessment and reassessments (blinded to the groups) and another who will apply the TFBM. Patients will be evaluated daily from day 1 (D1 - beginning of the chemotherapy cycle) until D10 or until healing of the lesions. The evaluation will consist of oral mucosa examination for grading of OM, pain assessment, quality of life, oral health, depressionand saliva evaluation of patients to assess. The analyses will be performed in the PASW 18.0 program, initially the evaluation of the data distribution will be performed by applying the Shapiro-Wilk and Kolmogorov-Smirnov tests. If, after applying these tests, the data show a normal distribution (p>0.05), the t-test will be used. If the distribution is non-normal after the application of the tests (p<0.05), the Wilcoxon test will be used. The p value will be set at 5%. Logistic regression will be used in adjusted models to estimate the probability of occurrence of OM.

DETAILED DESCRIPTION:
The main to compare two TFBM protocols using low-power laser and extraoral high-power laser in preventing OM in pediatric and adolescent oncology patients receiving treatment with antineoplastic chemotherapeutic agents. To evaluate the effectiveness of TFBM using extraoral low-power laser and high-power laser in the prevention and treatment of OM in pediatric patients receiving treatment with MTX-HD chemotherapy and its combinations.

Evaluate the impact of OM on the quality of life, anxiety, depression and pain of these patients. Evaluate the concentration of inflammatory and pro-inflammatory cytokines in saliva using the enzyme-linked immunosorbent assay (ELISA) in individuals undergoing chemotherapy who develop OM. Evaluate the role of NET and TSE in the saliva of patients undergoing chemotherapy who develop OM.

This is a controlled, randomized and blind clinical trial to evaluate the efficacy of the protocol using low-power and extraoral high-power TFBM in the prevention and treatment of OM in pediatric and adolescent oncology patients undergoing different chemotherapy protocols. The study will be conducted at the Hospital de Clínicas de Porto Alegre (HCPA) and AC. Camargo Center in the Pediatric Oncology Sector. After clarification and authorization of the responsible persons, they will have to sign the Informed Consent Form and the able research participants will sign the Informed Consent Form. The project will be registered in the Clinical Trials platform (https://clinicaltrials.gov/) and conducted according to the Consort checklist (Consolidated Standards of Reporting Trials). For data collection and management, the software REDcap® (Research Electronic Data Capture - Vanderbilt University, Nashville - Tennessee) and Google Drive will be used, where all forms regarding the evaluation of patients will be inserted.

A minimum of 34 pediatric and adolescent oncology patients diagnosed with malignancies, receiving intravenous (IV) QT of the following risk protocols for OM or some protocol that these chemotherapy drugs are included, will be included in this study, being: MTX-HD, combination chemotherapy of MTX-HD, doxorubicin and cyclophosphamide; and MTX-HD and cyclophosphamide. Patients who will be invited to participate in this study will be hospitalized for oncologic treatment and the informed consent form (ICF) and the informed consent form (ICF) will be applied at the Pediatric Oncology Department (3rd east) of the Hospital de Clínicas de Porto Alegre (HCPA). All patients included in this study will be submitted to a pre-treatment bedside dental evaluation and, if necessary, oral adaptation procedures (restorative, periodontal or tooth extraction needs) will be performed by the Hospital Dentistry of HCPA, and guidance will be given regarding the use of alcohol-based mouthwash, brushing with soft toothbrush and fluoride toothpaste, as well as guidance on the TFBM protocol and possible oral complications resulting from the QT treatment. All patients will be followed throughout the antineoplastic treatment, receiving reinforcement in oral hygiene orientation and guidance regarding side effects such as OM.

Information on gender (male/female), race, age (in years), medical history, underlying pathology and treatment modality (chemotherapy protocols used), pain medication used (medication category, dose and time of use), nutritional data (whether they are eating orally or using an esophageal tube) will be collected from the electronic medical records. One chemotherapy cycle from each patient included in the study will be evaluated.

in the study will be evaluated (MTX-HD, MTX-HD combined with cyclophosphamide and doxorubicin, and MTX-HD and cyclophosphamide). These data will be noted on a specific form for this study. If necessary, the evaluator will only have access to this form at the end of the patient's treatment in order to maintain the blinding of the study. atients will be randomly allocated into two groups: TFBMI (n = 17) and TFBME (n = 17). The study will be conducted by a dental surgeon who will perform the initial evaluation and reassessments (blinded to the experimental group) and another who will perform the TFBMT. Participants will be instructed not to give any spontaneous information about the treatment during the clinical evaluation, so that the treatment group to which they belong will not be identified. Following acceptance of participation in the study, the participants will go through a stratified randomization by chemotherapy protocol used in the treatment of childhood cancer.Randomization will be performed on Sealed Envelope software and participants will be allocated into 2 groups: Group I - TFBMI (n=17): Participants will receive TFBM from the first day of QT infusion, 5 times a week, from D1 (considered the beginning of chemotherapy infusion) until D10 (considered the peak of OM) in cases that the OM is maintained for longer the patients will be followed and treated until complete healing of the lesions.

Intraoral application: A low-power laser (Diode Semiconductor, Duo, MMOptics Ltda, São Carlos, SP, Brazil) with a wavelength of 660 nm (red) will be used, with an adaptation in power, since the MMOptics device with 40mW is no longer manufactured. Four anatomical areas will be irradiated perpendicularly in oral mucosa through several anatomical points with a distance of 1 cm approximately between them in order to cover the largest area per cm² in each region. Group II - TFBM with the extraoral high-power laser (n=17):

Participants will receive TFBM from the first day of QT infusion, 5 times a week, from D1 (considered the beginning of chemotherapy infusion) until D10 (considered the peak of OM) in cases that the OM remains longer the patients will be followed and treated until complete healing of the lesions.

A gallium-aluminum arsenide diode laser (Gemini® manufactured by Azena Medical, LLC, distributed by Ultradent Products, Inc.) with double wavelength 810 + 980 nm, previously standardized and calibrated for extraoral application by power meter (Coherent Inc, Santa Clara, CA) will be used. The equipment will be programmed with 1 W of power. The responsible researcher will execute the TFBM and he will not carry out any type of evaluation.

The application of the questionnaires and clinical evaluation will be carried out by another examiner who will not be aware of the group to which each patient is allocated.

During the QT period, all patients will be evaluated daily for the presence and grading of OM and pain. Saliva samples will be collected from participants of all groups, in three moments of clinical evaluation, for further analysis of inflammatory cytones, NET and TSE.

Questionnaires about quality of life, childhood depression and perception of parents and guardians on the quality of life of patients will be carried out.

Initially, the evaluation of data distribution will be carried out from the application of the Shapiro-Wilk and Kolmogorov-Smirnov tests. If from the application of these tests, the data show normal distribution (p>0.05), the test will be used t. If the distribution proves to be non-normal after applying the tests (p<0.05), the Wilcoxon test will be used. The p-value will be set to 5%. Logistic regression will be used in adjusted models to estimate the probability of occurrence of mucositis (dependent variable) in relation to clinical and demographic variables (independent variables). Analyzes will be performed using the PASW 18.0.3.11 program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant neoplasia (hematological or solid tumors);
* Responsible and participants agree to the study participation after reading and signing the Informed Consent Form (ICF) and Informed Term of Consent (TALE) for participation in Clinical Research;
* They performed the chemotherapy infusions hospitalized in the pediatric oncology department of the 3rd east of HCPA;
* Received the following chemotherapy protocols: MTX-HD, combination chemotherapy of MTX-HD, doxorubicin and cyclophosphamide; and MTX-HD and cyclophosphamide.

Exclusion Criteria:

* Participants will be excluded who:
* Patients over the age of 18 years
* Patients who will undergo HSCT

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis evalution according World Health Organization (WHO) scale | 16 months
  According to the classification criteria to World Health Organization (WHO, 1979): Grade 0 None Grade 1 Erythema, oral mucosal tenderness, pain Grade 2 Erythema, ulcerated lesion, can swallow solid food Grade 3 Ulcerated lesions require only liquid diet Grade 4 Impossible to eat, solid or liquid
Oral mucositis evalution according National Cancer Institute (NCI) scale | 16 months
  According to the classification criteria to NCI 1999: Grade 0 None Grade 1 Painless ulcers, erythema or mild pain in the absence of lesions Grade 2 Painful erythema, edema or ulcers but can eat/swallow Grade 3 Painful erythema, edema or ulcers requiring IV hydration Grade 4 Severe ulcerations or requires parenteral/enteral nutrition support or prophylactic intubation
Oral mucositis Children's International Mucositis Evaluation Scale (CHIMES) | 16 months
  Childhood Mucositis Evaluation (CHIMES). For the CHIMES- BR version items 1-4 are scored from 0 (best score) to 5 (worst score), the remaining items are answered with yes or no response and are assigned scores of 0 and 1, respectively. The maximum total score is 23.

SECONDARY OUTCOMES:
Pain evalution The Visual Analogic Scale (VAS) | 16 months
  The child will be asked to choose the face that best describes how he feels. The VAS will be represented by a 10 cm straight line where 0 corresponds to the best situation and 10 to the worst situation. The research participants will be instructed by the evaluator to mark a point on the 10 cm line
Pain evolution - Wong Baker Faces | 16 months
  For the Wong-Baker faces scale it will be explained to the children that each face represents a person who is happy because they have no pain, or sad because they have a little or a lot of pain. Face O is very happy because he has no pain. Face 1 has only a little pain. Face 2 has a little more pain. Face 3 has even more pain. Face 4 has a lot of pain. Face 5 has maximum pain, although it does not always provoke crying.
Quality of Life Assessment | 16 months
  Oral Health Impact Profile (OHIP-14) will also be used as a questionnaire to assess patients' quality of life in relation to oral health. OHIP-14 summarizes the following seven domains of impact on daily activities as a result of oral problems: limitation (domain 1), physical pain (domain 2), discomfort (domain 3), physical activity (domain 4), psychological impairment (domain 5), social impairment (domain 6), and disability (domain 7). The OHIP-14 instrument consists of 14 questions related to oral health, with five response options: 0 = never, 1 = almost never, 2 = occasionally, 3 = quite often, 4 = very often.
Caregivers' Quality of Life Assessment | 16 months
  Parental-caregiver perceptions questionnaire (P-CPQ), short version will be used, which has 13 questions divided into three domains: oral symptoms (3 items), functional limitations (4 items) and emotional well-being (6 items). The items refer to the frequency of events related to oral health in the last three months. Each question has 5 response options: (0) never, (1) once or twice, (2) sometimes, (3) frequently, (4) every day or almost every day. The total score ranges from 0 to 52 points. The answer with "don't know" is also an option that can be selected, and is measured with a value of zero. Higher values indicate a more negative perception by the mother/father/caregiver regarding the impact of oral conditions on the quality of life of their children. Scores for each of the three domains are also possible. The child's oral health and general well-being are also recorded on the instrument, using a five-point response format from "excellent" to "bad" for oral
Anxiety and depression assessment | 16 months
  The Children's Depression Inventory (CDI) has 27 questions regarding depressive symptoms in children and adolescents. Each question has three response options in different contexts for clinical applicability, especially diagnosis of depression and anxiety traits (KOVACS, 1985).
Analysis cytokines | 16 months
  The collection of non-stimulated saliva is performed in an environment with artificial light, with the patient sitting with eyes open, head slightly tilted down, without speaking, opening the mouth or swallowing saliva during the moment of collection, before clinical care. All the saliva produced, within a 5-minute interval, is collected in a sterile millimeter Falcon tube that will be handed over by the researcher at the time of collection. The collections will be made in 3 moments (D1, D7 and at the end of the chemotherapy cycle) for later analysis of cytokines, ELISA will be used to quantify the levels of inflammatory and pro-inflammatory cytokines in the saliva will be evaluated the cytokines IL-2, IL- 6, IL-8, IL-10, IL-β and TNF-F.
Analysis NET and TSE | 16 months
  The saliva collections will be made in 3 moments (D1, D7 and at the end of the chemotherapy cycle) for later analysis of the NET and TSE. For the quantification of NET in saliva, the anti-MPO antibody and the DNA quantification kit PicoGreen® dsDNA Assay Kit (Invitrogen, USA) will be used. Co-localization of extracellular DNA with histones, neutrophil elastase and myeloperoxidase will confirm the classic characteristics of NETs and will be determined by spectrofluorometric analysis (excitation at 484 nm and emission at 520 nm) in an automated reader. For the quantification of TSE in saliva, the anti-MBP Ab antibody (clone AHE-2, BD Pharmingen) and the DNA quantification kit PicoGreen® dsDNA Assay Kit (Invitrogen, USA) will be used. The granules will be confirmed by spectrofluorometric analysis (484nm excitation and 520nm emission) in an automated reader. Saliva collection does not cause discomfort or harm to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Manoela D Martins, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Fabio A Alves, PhD, Study Chair — A.C Camargo Center
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the outcomes, for one year
Access Criteria: If formally solicited and referencead by the researcher interestend